CLINICAL TRIAL: NCT02154165
Title: Comparison Between Turquoise and Blue Light in Treatment of Neonatal Jaundice Using Light Emission Diodes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Principal Investigator, Helene Nørrelund, MD, University of Aarhus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PKV 2013
Record Dates: First submitted 2014-05-30; First posted 2014-06-03 (Estimated); Last update posted 2014-06-03 (Estimated); Status verified 2014-05

CONDITIONS: Uncomplicated Neonatal Hyperbilirubinemia
Keywords: Neonatal hyperbilirubinemia; Phototherapy; Light emitting diodes; Blue light; Turquoise light
MeSH Terms: conditions — Hyperbilirubinemia, Neonatal | interventions — Phototherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Blue light wavelenght 460 nm (Active Comparator)
  Interventions: Other: Phototherapy
- Turquoise light wavelength 499 nm (Active Comparator)
  Interventions: Other: Phototherapy

INTERVENTIONS:
Other: Phototherapy — The infants were randomized to phototherapy with either blue og turquoise light

SUMMARY:
The optimal wavelength for phototherapy for neonatal jaundice remains to be clarified by clinical studies. Previous iv vivo studies have shown that turquoise light at wavelength about 490 nm is more efficacious than blue light at wavelength 460 nm, which is the golden standard in phototherapy treatment today. Though, previous studies used light tubes, today we use light emitting diodes (LED'S).

The overall aim of this study was therefore to compare the efficacy of turquoise LED's versus blue LED's for decreasing total serum bilirubin in neonates with gestational age > 33 weeks and uncomplicated hyperbilirubinemia.

ELIGIBILITY:
Inclusion Criteria:

* Newborns with gestational age >33 weeks and neonatal hyperbilirubinemia requiring treatment with phototherapy according to the national guidelines

Exclusion Criteria:

* Haemolytic disease (Rhesus and Kell blood type isoimmunization, spherocytosis)
* Liver disease

Min Age: 33 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2013-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Decrease in total serum bilirubin | 24 hours
  The infants were treated with phototherapy for 24 hours, which is the standard treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Neonatal department, Aalborg University Hospital, Aalborg, Denmark